CLINICAL TRIAL: NCT06349798
Title: Early and Late Effects of Nefopam in Multimodal Analgesia After Total Hip Arthroplasty (NEFARTHRO): a Multicentric Randomized Controlled Trial.
Brief Title: Early and Late Effects of Nefopam in Multimodal Analgesia After Total Hip Arthroplasty (NEFARTHRO)
Acronym: NEFARTHRO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DR200177
Record Dates: First submitted 2024-01-23; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Total Hip Arthroplasty
MeSH Terms: interventions — Nefopam; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Multicenter, double-blind, randomized controlled trial in 3 parallel groups (placebo group, nefopam bolus group and nefopam Continuous Intra-Venous Infusion CIVI group).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patient, investigator and outcome assessor will be blind., A nurse anesthetist who will not be involved in the follow up of the patient will receive the kit and prepare the syringes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nefopam "bolus" group (Experimental)
  Interventions: Drug: Nefopam
- Nefopam "CIVI" group (Experimental)
  Interventions: Drug: Nefopam
- Control group (Placebo Comparator)
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Nefopam — 20 mg nefopam in 50 ml of saline, during a 30 min infusion, before end of procedure, then a similer bolus every 4 h for 24 h (6 injections in total) + continuous intravenous infusion of placebo (2 mL/h saline)
  Arms: Nefopam "bolus" group
Drug: Nefopam — 20 mg nefopam in 50 ml of saline, during a 30 min infusion, before end of procedure, then a bolus of placebo every 4 h for 24 h (6 injections in total) + continuous infusion of 100 mg nefopam over 24 h (in 48 mL saline, 2 mL/h)
  Arms: Nefopam "CIVI" group
Drug: NaCl 0.9% — 50 ml of saline, during a 30 min infusion, before end of procedure, followed by a bolus of placebo every 4 hours for 24 hours (6 injections in all) + continuous infusion of placebo (2 mL/h of physiological saline)
  Arms: Control group

SUMMARY:
NEFARTHRO is a multicentric randomized controlled trial comparing the effects of discontinuous infusions of nefopam (bolus) versus continuous infusion of intravenous nefopam (via an infusion pump) versus placebo on the opioid-request during the first 24 hours following a Total Hip arthroplasty, as part of multimodal analgesia including at least paracetamol and a Non-Steroidal Anti-Inflammatory Drug (NSAID).

The primary endpoint is cumulative morphine consumption for the first postoperative 24 hours, expressed in mg of iv equivalent morphine, including titration in the Post Anesthesia Care Unit (PACU).

Patients will be followed during 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years, fluent in French.
* Planned primary or secondary total hip replacement, regardless of surgical approach or type of prosthesis.
* Receiving paracetamol and ketoprofen postoperatively.
* Under general anesthesia or spinal anesthesia (without intrathecal morphine).
* Participant affiliated to a social security scheme
* Participant's free, informed and written consent

Exclusion Criteria:

* Septic or carcinological surgery
* Allergy to paracetamol, nefopam or NSAIDs
* Angle-closure glaucoma
* Prostate adenoma
* history of convulsion
* Nocturnal pollakiuria in men with more than two risings per night
* Severe hepatic (Child C) or cardiac insufficiency (LVEF < 30%)
* Renal insufficiency with creatinine clearance < 50 mL/ min according to Cockroft's formula
* Active peptic ulcer or history of digestive bleeding or peptic perforation
* Patients with opioid treatment for chronic pain other than coxarthrosis (fentanyl, oral morphine > 50mg/d or equivalent)
* Protected patient: safeguard of justice, guardianship or curatorship
* Incomprehension or inability to use a numerical rating scale or to self-assess/manage pain
* Pregnancy or breast-feeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Cumulative morphine consumption from the end of surgery (Day 0 - Hour 0) to the first 24 hours after surgery, expressed in mg of intravenous morphine (including titration in the Post-Anesthesia care Unit PACU). | between Day 0 - Hour 0 and Hour 24 post surgery

SECONDARY OUTCOMES:
Maximum self-assessed pain using the Numeric Rating Scale ranging from 0 (no pain) to 10 (maximum pain) at rest in the PACU, at rest and on walking between PACU discharge and Hour 24, at Hour 24, and at hospital discharge. | at PACU, between PACU discharge and Hour 24, at Hour 24 and at Day 5 of hospital discharge
Time to return to walking. | At Hour 24, at Day 5 or at discharge, whichever came first and at Month 6
Time to leave room. | At Hour 24, at Day 5 or at discharge, whichever came first and at Month 6
Time to climb stairs. | At Hour 24, at Day 5 or at discharge, whichever came first and at Month 6
Length of stay. | At Day 0 - Hour 0 up to Day 5 or at discharge
Time to abandon canes/crutches. | At Hour 24, at Day 5 or at discharge, whichever came first and at Month 6
Opioid analgesic consumption between days 1 and 5 or at hospital discharge | at Hour 24 and up to day 5
Chronic pain at 6 months (at rest and walking) using a standardized phone questionnaire. | At Month 6
Neuropathic pain score (DN2)The DN2 is a simplified version of the DN4, with 7 items: burning, painful cold, electric shocks, tingling, pins and needles, numbness, itching (scored 0=absent, 1=present). | At Hour 24 and Month 6
Incidence of all serious AEs during patient follow-up and non-serious AEs. | at Hour 24 and up to day 5
Incidence of patients with morphine side effects | at Hour 24 and up to day 5
  Incidence of patients with morphine side effects: nausea, vomiting, use of anti-nausea medication, pruritus requiring modification of management, urinary retention, use of urinary antispasmodics or urethral catheterization/suprapubic catheter, or abnormal drowsiness.
Financial impact of spreading the recommended strategy following the results of the clinical study, estimated per year and over a 5-year period, from the point of view of the French Health Insurance and from the hospital perspective. | 5 years
  These financial impacts will be estimated using budget impact models.

CONTACTS AND LOCATIONS:
Overall Officials: Francis REMERAND, MD PhD, Principal Investigator — CHRU de Tours
Locations (7):
- France (7):
  - Anaesthesia - Intensive care, Angers
  - Anaesthesia - Intensive care, Blois
  - Anaesthesia - Intensive care, Chartres
  - Anaesthesia - Intensive care, Nantes
  - Anaesthesia - Intensive care, Orléans
  - Anaesthesia - Intensive care, Poitiers
  - Anesthesia - intensive care, Tours

IPD SHARING:
Plan to Share IPD: No